CLINICAL TRIAL: NCT01360008
Title: FREEZE Cohort Study
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: FREEZE
Record Dates: First submitted 2011-05-13; First posted 2011-05-25 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2017-09

CONDITIONS: Arrhythmia
Keywords: Cardiac arrhythmia; Catheter ablation; Cohort Study; cryoballoon; radiofrequency
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cryo ablation: Patients with first Ablation of atrial fibrillation treated by cryo ablation
- RF ablation: Patients with first Ablation of atrial fibrillation treated by Radio frequency ablation

SUMMARY:
Safety and efficacy in radiofrequency (RF) or cryoballoon atrial fibrillation (AF) ablation will be investigated in a cohort study design in experienced electrophysiologic (EP) centers analyzing propensity-matched cohorts.

DETAILED DESCRIPTION:
Prior to participation in the cohort-study each EP center had to perform a minimum of 50 RF or 50 cryoballoon approaches. To insure the consecutiveness of recruitment, participating centers have to announce the intention to ablate the patient prior to the procedure to the coordinating center in Ludwigshafen. After inclusion of 500 patients with well accepted criteria for AF ablation undergoing cryoballoon pulmonary vein isolation (PVI) in experienced german EP centers inclusion of patients will be extended to european centers. A total of 4.000 patients will be included in the cohort-study, 2.000 in both the cryoballoon and the RF arm.

ELIGIBILITY:
Inclusion Criteria:

* Documented paroxysmal AF (2 episodes of PAF within the last 3 months) or Persistent AF (lasting < 1 year)
* First ablation of AF
* Age ≥18 years
* Documented inefficacy of at least 1 AAD not including β-blockers
* Written informed consent

Exclusion Criteria:

* Longstanding persistent AF lasting > 1 year
* Acute coronary syndrome (ACS)
* Heart failure NYHA IV
* Thrombocytosis, thrombocytopenia
* Any condition contraindicating chronic anticoagulation
* Stroke or TIA within 6 months prior to ablation
* Uncontrolled hyperthyroidism
* Pregnancy
* Life expectancy < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AF ablation targeting
Sampling Method: Non-Probability Sample
Enrollment: 4071 (Actual)
Dates: Start 2011-04; Primary Completion 2016-01 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
AF recurrency rate (any detected episode lasting > 30 sec) at 12 months follow up | Admission to hospital until 12 months thereafter

SECONDARY OUTCOMES:
Comparison of complication rates (any complications and major complications) at 12 months follow-up | Admission to hospital until 12 months thereafter
Specific complication aspects with respect to phrenic nerve palsy and PV stenosis | Admission to Hospital until 12 months thereafter
Efficacy (AF recurrency rates), safety (complication rates), and procedural parameters in cryoballoon or RF ablation as means for assessing advantages of preprocedural CT or MRI scan performing 3 D anatomy of the left atrium and pulmonary veins | Admission to Hospital until 12 months thereafter
Persistent AF: Impact on efficacy analyzing procedural aspects in cryoballoon PVI | Admission to Hospital until 12 months thereafter
Real-time ECG-monitoring of PV-isolation during freezing: Does the microcircular mapping catheter add significant benefit to the cryoballoon procedure | Admission to Hospital until 12 months thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Hoffmann, MD, Principal Investigator — Klinikum Bogenhausen, München
Locations (37):
- Mission Hospital, Inc., Asheville, North Carolina, United States
- Allgemeines KH Linz, Linz, Austria
- Germany (30):
  - Klinikum Aschaffenburg, Aschaffenburg
  - Herz-Zentrum Bad Krozingen, Bad Krozingen
  - Kerckhoff-Klinik, Bad Nauheim
  - Herz- und Gefäßklinik Bad Neustadt; Klinik für Kardiologie II, Bad Neustadt an der Saale
  - Herz- und Diabeteszentrum, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin (Kardiologie), Berlin
  - Vivantes Klinikum Am Urban, Berlin
  - Klinikum Bielelfeld - Klinik für Kardiologie und internistische Intensivmedizin, Bielefeld
  - Universitätsklinikum Bonn (Med. Klinik und Poliklinik II), Bonn
  - Klinikum Coburg, Coburg
  - St. Vinzenz Hospital Köln-Nippes, Cologne
  - Praxisklinik Herz und Gefäße, Dresden
  - Elisabeth-Krankenhaus Essen; Klinik für Kardiologie und Angiologie, Essen
  - Städt. Klinikum Frankfurt Höchst, Frankfurt
  - Cardioangiologisches Centrum Bethanien - CCB, Frankfurt
  - Universitäres Herzzentrum Eppendorf, Hamburg
  - Asklepios Klinik St. Georg, Hamburg
  - Universitäres Herzzentrum, Hamburg
  - Klinikum Siloah, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Städt. Klinikum Hildesheim, Hildesheim
  - Klinikum Ingolstadt, Ingolstadt
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Universitätsklinik Schleswig-Holstein Campus Lübeck, Lübeck
  - Universitätsmedizin Mainz, Mainz
  - Isar Herzzentrum München, München
  - Krankenhaus München Bogenhausen, München
  - Universitätsklinikum Münster, Münster
  - Klinikum Traunstein, Traunstein
  - Schwarzwald-Baar-Klinikum Villingen-Schwenningen GmbH, Villingen-Schwenningen
- Evangelismos General Hospital, Athens, Greece
- South Africa (3):
  - Sunninghill Hospital, Johannesburg
  - Panorama Medi-Clinic, Panorama
  - Milpark Hospital, Parktown West
- University Hospital Virgen de la Arrixaca, El Palmar - Murcia, Spain

IPD SHARING:
Plan to Share IPD: No
De-identified patient data will be published after end of follow up period

REFERENCES:
- [Derived] Pongratz J, Kuniss M, Wu L, Tebbenjohanns J, Nolker G, Dorwarth U, Kuck KH, Jochen S, Hoffmann E, Straube F; FREEZE Cohort Study Investigators. Impact of intracardiac echocardiography usage on the safety of cryoballoon atrial fibrillation ablation: Subanalysis of the prospective FREEZE cluster cohort study. J Cardiovasc Electrophysiol. 2023 Oct;34(10):2029-2039. doi: 10.1111/jce.16060. Epub 2023 Sep 8. PMID 37681996
- [Derived] Metzner A, Straube F, Tilz RR, Kuniss M, Noelker G, Tebbenjohanns J, Andresen D, Wieneke H, Stellbrink C, Franke J, Dorwarth U, Carion PL, Holbrook R, Hochadel M, Senges J, Hoffmann E, Kuck KH; FREEZE Cohort Study Investigators. Electrophysiology lab efficiency comparison between cryoballoon and point-by-point radiofrequency ablation: a German sub-analysis of the FREEZE Cohort study. BMC Cardiovasc Disord. 2023 Jan 9;23(1):8. doi: 10.1186/s12872-022-03015-8. PMID 36624380
- [Derived] Hoffmann E, Straube F, Wegscheider K, Kuniss M, Andresen D, Wu LQ, Tebbenjohanns J, Noelker G, Tilz RR, Chun JKR, Franke A, Stellbrink C, Garcia-Alberola A, Dorwarth U, Metzner A, Ouarrak T, Brachmann J, Kuck KH, Senges J; FREEZE Cohort Study Investigators. Outcomes of cryoballoon or radiofrequency ablation in symptomatic paroxysmal or persistent atrial fibrillation. Europace. 2019 Sep 1;21(9):1313-1324. doi: 10.1093/europace/euz155. PMID 31199860
- [Derived] Straube F, Dorwarth U, Ammar-Busch S, Peter T, Noelker G, Massa T, Kuniss M, Ewertsen NC, Chun KR, Tebbenjohanns J, Tilz R, Kuck KH, Ouarrak T, Senges J, Hoffmann E; FREEZE Cohort Investigators. First-line catheter ablation of paroxysmal atrial fibrillation: outcome of radiofrequency vs. cryoballoon pulmonary vein isolation. Europace. 2016 Mar;18(3):368-75. doi: 10.1093/europace/euv271. Epub 2015 Oct 25. PMID 26504108
- [Derived] Straube F, Dorwarth U, Vogt J, Kuniss M, Heinz Kuck K, Tebbenjohanns J, Garcia Alberola A, Chun KR, Souza JJ, Ouarrak T, Senges J, Brachmann J, Lewalter T, Hoffmann E. Differences of two cryoballoon generations: insights from the prospective multicentre, multinational FREEZE Cohort Substudy. Europace. 2014 Oct;16(10):1434-42. doi: 10.1093/europace/euu162. Epub 2014 Jul 3. PMID 24994074